CLINICAL TRIAL: NCT05273684
Title: High-intensity Interval Training in Patients With COPD: a Fidelity and Tolerability Study
Acronym: COPDEX-HIIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Ronan Berg, MD, DMSc, Associate professor, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CFAS_2021_1
Record Dates: First submitted 2021-11-09; First posted 2022-03-10 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: COPD
Keywords: HIIT; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 4*4 followed by 10*1 or 10*1 followed by 4*4 (Experimental): Following baseline measurements, participants are allocated to the random sequence, by which they will complete the two HIIT protocols ⟨http://www.randomization.com⟩ and based on this, patients are randomized to a specific testing sequence.
  Interventions: Other: High intensity interval training

INTERVENTIONS:
Other: High intensity interval training — Participants will undergo 4x4 and 1x10 minutes of interval training on two separate days.

SUMMARY:
Although high-intensity training (HIIT) is widely used in the rehabilitation of patients with chronic obstructive pulmonary disease (COPD), the optimal duration of intervals in terms of patient tolerability and fidelity is unknown.Thus, we will examine the fidelity and tolerability of the two most commonly used HIIT protocols, the classical so-called 4x4min vs. 10x1min in patients with moderate to severe COPD.

DETAILED DESCRIPTION:
12 patients with severe to moderate COPD will be included in the study, where two different HIIT interventions will be compared with regards to fidelity and tolerability. Baseline measurements will be performed to assess fitness and cardiopulmonary health status for the included patients. The baseline measurements include a medical health interview and examination (blood pressure, heart rate, ECG), a maximal oxygen consumption (VO2max) test, lung function testing (dynamic spirometry, whole body plethysmography, diffusing capacity), and an assessment of body composition. The following two visits consist of two different HIIT protocols.

Each training session is evaluated by Borg Scale (5) and the Likert Scale (6), as well as time spent in with a heart rate above 85% of maximum. Each HIIT session is separated by at least a 3-day wash-out period.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* 18-80 years
* Moderate to severe COPD(GOLD stage II to III)

Exclusion Criteria:

* Known ischaemic heart disease
* Known heart failure
* Previous or current coronavirus disease 2019 (COVID-19)
* Dementia or other severe neurological disease
* Known vascular
* Symptoms of disease within 2 weeks prior to the study
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Exercise feasibility: Relative dose intensity (RDI) of exercise | 1 week
  RDI (%) of exercise, defined as prescribed exercise dose / performed exercise dose x 100
  Evaluated with a Red-Amber-Green system:
  * Green: If ≥85% of the training is completed
  * Amber: If 50-85% of the training is completed
  * Red: If ≤ 50% of the training is completed
Exercise feasibility: Exercise sessions requiring dose modifications | 1 week
  Incidence of exercise sessions requiring dose modifications, defined as any deviation from the prescribed exercise.
Exercise tolerability: Subjective rating of the exercise session | 1 week
  Tolerability is measured with a 10-point Likert scale, where the participants evaluate the two HIIT protocols.
  They will anser two quesitens:
  1. How tolerable was todays traning?
  2. How much did you enjoy todays training? Where 1 means not at all, and 10 means alot.
  The Likert scale is scored as:
  Red: 1-2 Amber: 3-4 Green: +5
Exercise feasibility: Exercise sessions attendance rate | 1 week
  Exercise sessions attendance rate (%), defined as number of attended exercise sessions / number of prescribed exercise sessions x 100

CONTACTS AND LOCATIONS:
Overall Officials: Ronan Berg, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nymand SB, Hartmann J, Rasmussen IE, Iepsen UW, Ried-Larsen M, Christensen RH, Berg RMG. Fidelity and tolerability of two high-intensity interval training protocols in patients with COPD: a randomised cross-over pilot study. BMJ Open Sport Exerc Med. 2023 Mar 8;9(1):e001486. doi: 10.1136/bmjsem-2022-001486. eCollection 2023. PMID 36919122